CLINICAL TRIAL: NCT03283826
Title: A Phase 1/2, Two-part, Open-label Dose-escalation and Double-blind, Placebo-controlled Dose-expansion Study With an Open-label Extension to Evaluate the Safety and Efficacy of ATA188 in Subjects With Progressive Multiple Sclerosis
Brief Title: Phase 1/2 Study to Evaluate the Safety and Efficacy of ATA188 in Subjects With Progressive Multiple Sclerosis
Acronym: EMBOLD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated as primary endpoint was not achieved
Sponsor: Atara Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ATA188-MS-101; NCT03283826 (Registry Identifier: Clinicaltrials.gov)
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Primary Progressive Multiple Sclerosis; Secondary Progressive Multiple Sclerosis
Keywords: Multiple Sclerosis (MS); Primary Progressive Multiple Sclerosis; Secondary Progressive Multiple Sclerosis; Epstein-Barr Virus (EBV); EBV-associated Multiple Sclerosis; Inflammation; Central Nervous System; Autoimmune Disease; Autoimmunity; Demyelination; Cell Therapy; T-cell; Allogeneic; EBV viremia; Off-the-shelf (T cells)
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis; Epstein-Barr Virus Infections; Inflammation; Autoimmune Diseases; Demyelinating Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATA188 (Experimental): Participants in Parts 1 and 2 will receive ATA188 intravenously as described in the Detailed Description.
  Interventions: Biological: ATA188
- Placebo (Placebo Comparator): Participants in Part 2 will receive placebo matching to ATA188 intravenously as described in the Detailed Description (i.e., will receive placebo only in the first year, and thereafter will receive ATA188 for the remainder of the study).
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: ATA188 — ATA188 is being investigated as an off-the-shelf, allogeneic T-cell immunotherapy for the treatment of EBV+ progressive multiple sclerosis.
  Other Names: Epstein-Barr Virus-directed cytotoxic T lymphocytes (CTLs); EBV-CTLs; EBV-targeted T-cell
  Arms: ATA188
Drug: Placebo — Placebo matching to ATA188
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of ATA188 as a monotherapy in Parts 1 and 2, to determine the recommended Part 2 dose (RP2D) of ATA188 as monotherapy in Part 1, and to evaluate the effect of ATA188 treatment on clinical disability, as assessed by confirmed Expanded Disability Status Scale (EDSS) improvement at 12 months in Part 2 in participants with progressive forms of multiple sclerosis (MS) (primary progressive multiple sclerosis [PPMS] and secondary progressive multiple sclerosis [SPMS]).

DETAILED DESCRIPTION:
This is a multicenter, 2 part study in adult participants with progressive forms of MS (PPMS/SPMS) with an open-label, single-arm, sequential dose-escalation period (Part 1) and a double-blind, randomized, placebo-controlled dose-expansion period (Part 2) followed by open-label extension (OLE) period. Part 2 and the OLE have been initiated by the sponsor's discretion based on a review of data from the dose-escalation cohorts.

This study will evaluate the safety and efficacy of ATA188 administered by intravenous (IV) infusion. ATA188 will be selected for each participant based on matching 2 or more human leukocyte antigen (HLA) alleles shared between ATA188 and the participant, at least 1 of which is a HLA-restricting allele.

In Part 1, participants received 2 cycles of ATA188 and entered 12 months follow-up period after the last dose of ATA188. Participants who completed at least the first year of the dose-escalation period and were active in the study have entered the OLE period. In OLE period, participants will receive the same RP2D assigned to Part 2 participants at the time of the Part 1 participant's first dose in each year of the OLE. In OLE period, participants will receive 1 cycle of ATA188 treatment every 12 months (Q12M) for up to 4 years (ie, Years 2 to 5). Otherwise, end of study (EOS) visit will be conducted at 24 months after Cycle 1 Day 1.

In Part 2, participants will be randomized in 1:1 ratio to receive ATA188 at the RP2D or matching placebo, stratified by progressive MS diagnosis (PPMS vs SPMS) and any prior exposure to anti-CD20 therapy (yes vs no). Participants will receive 2 cycles of ATA188 at the RP2D or matching placebo and will be followed for at least 12 months after the first dose of study drug (ie, Year 1). In second year (Year 2), participants who received placebo in Year 1 will receive 2 cycles of ATA188 at the RP2D assigned at randomization and participants who received ATA188 at the RP2D in Year 1 will receive 1 cycle of ATA188 (at the RP2D assigned at randomization) and 1 cycle of placebo to maintain the blind. Participants who complete Year 2 will enter the OLE period to receive ATA188 Q12M for up to 3 years (ie, Years 3 to 5) at the RP2D that was last selected by the sponsor for Part 2. The end of study visit will be scheduled at 5 years (60 months) after the first dose of study drug (ie, Cycle 1 Day 1).

Based on interim analysis, the recruitment for Parts 1and 2 have completed.

ELIGIBILITY:
Inclusion Criteria:

* For Part 1: History of progressive forms of MS (PPMS or SPMS), as defined by the 2010 Revised McDonald criteria for the diagnosis of MS
* For Part 1: 18 to < 66 years of age
* For Part 1: EDSS scores of 3.0 to 7.0. Participants with EDSS scores of 6.5 to 7.0 must retain measurable upper limb function as assessed by the 9-hole Peg Test (9HPT).
* For Part 2: Current diagnosis of a progressive form of MS (PPMS or SPMS) as defined by the 2017 Revised McDonald criteria
* For Part 2:18 to < 61 years of age
* For Part 2:EDSS scores of 3.0 to 6.5
* Positive EBV serology
* Willing and able to provide written informed consent

Exclusion Criteria:

* Clinical relapse as follows: For Part 1: Active clinical relapse between providing informed consent and the first dose of study drug. For Part 2: Documented clinical and/or radiological relapse for 2 years prior to screening, including gadolinium (Gd)-enhancing lesion(s) on any brain MRI scans available during this period (A participant will also be considered ineligible if any clinical and/or radiological relapse is reported between screening and the first dose of study drug.)
* Concurrent serious uncontrolled or unresolved medical condition, such as infection, limiting protocol compliance or exposing the subject to unacceptable risk
* Positive serology and/or nucleic acid testing (NAT) for human immunodeficiency virus (HIV), active hepatitis B virus (HBV) infection or carrier status for HBV, active hepatitis C virus (HCV) infection
* For Part 1: Positive serology for syphilis or human T cell lymphotrophic virus I/II
* Uncontrolled psychosis, uncontrolled depression or suicide risk, substance dependence, or any other psychiatric condition that may compromise the ability to participate in this trial
* Clinically significant abnormalities of full blood count, renal function, or hepatic function
* Any contraindication to MRI and/or Gd, eg., any object that is reactive to strong static magnetic, pulsed-gradient fields including any metallic fragments or foreign body (eg, aneurysm clip[s], pacemakers, electronic implants, shunts)
* Any history of cancer (as exceptions, successfully treated non-melanoma skin cancer or carcinoma in situ of the cervix with a < 5% chance of recurrence within 12 months of providing informed consent are allowed.)
* Prior therapy with corticosteroids (within 2 weeks before Cycle 1 Day 1)
* Prior therapy (30 days) B-cell depleting agent (eg, anti-CD20 agents such as ocrelizumab); participant must be progressing despite therapy to be eligible
* For Part 1: Prior therapy (6 half-lives or 30 days whichever is longer) with cladribine, glatiramer acetate, interferon β, dimethyl fumarate, methotrexate, azathioprine, cyclosporine, fingolimod, natalizumab, teriflunomide, mitoxantrone, cyclophosphamide, any other immunosuppressant or cytotoxic therapy (other than steroids), antithymocyte globulin or similar anti-T-cell antibody therapy, or any other investigational product
* For Part 1: Any previous treatment with alemtuzumab, ablative stem cell transplant, or EBV T-cell therapy
* For Part 2: Prior therapy (6 half-lives or 30 days whichever is longer) with IV immunoglobin, plasmapheresis, Bruton's tyrosine kinase inhibitors, all sphingosine 1-phosphate receptor modulators (eg, fingolimod), glatiramer acetate, interferon β, nuclear factor (erythroid-derived 2)-like 2 (Nrf2) activators (eg, dimethyl fumarate), methotrexate, azathioprine, cyclosporine, natalizumab, teriflunomide, mitoxantrone, cyclophosphamide, any other immunosuppressant or cytotoxic therapy (other than steroids), antithymocyte globulin or similar anti-T-cell antibody therapy, or any other investigational product
* For Part 2: Any previous treatment with cladribine, alemtuzumab, ablative stem cell transplant, or EBV T-cell therapy
* Unresolved reactions from previous therapies that may, in the investigator's opinion, impact the safety of the participant or the conduct of this study
* Unwilling to use protocol specified contraceptive methods
* Women who are breastfeeding
* Pregnancy
* Inability or unwillingness to comply with study procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Part 1: Incidence of adverse events | At 12 months after the first dose of study drug
Part 1: Incidence of clinically significant changes in laboratory tests, electrocardiograms (ECGs), and vital signs | At 12 months after the first dose of study drug
Part 1: Recommended Part 2 dose of ATA188 monotherapy | Day 1 to Day 35 of Cycle 1 for each participant in dose escalation part (approximately 1 year)
Part 2: Percentage of participants with confirmed expanded disability status scale (EDSS) improvement at 12 months | At 12 months after the first dose of study drug

SECONDARY OUTCOMES:
Part 1: Change from baseline in EDSS score | At 12 months after the first dose of study drug
Part 2: Percentage of participants with confirmed EDSS improvement at 15 months | At 15 months after the first dose of study drug
Part 2: Percentage of participants with sustained disability improvement (SDI; ie, confirmed EDSS improvement or 20% decrease in timed 25-foot walk [T25W]) at 12 months | At 12 months after the first dose of study drug
Part 2: Percentage of participants with SDI at 15 months | At 15 months after the first dose of study drug
Part 2: Change from baseline in immunoglobulin G (IgG) index | At 9 months after the first dose of study drug

OTHER OUTCOMES:
Change from baseline in cervical spinal cord volume on MRI scans | At 12 months after the first dose of study drug
Change from baseline in whole brain volume on MRI scans | At 12 months after the first dose of study drug
Change from baseline in number of Gd-enhancing and new or enlarging T2 lesions on brain MRI scans | At 12 months after the first dose of study drug
Change from baseline in IgG production | At 12 months after the first dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Kiren Kresa-Reahl, MD, Study Director — Atara Biotherapeutics
Locations (31):
- United States (25):
  - University of California, San Diego, La Jolla, California
  - Kaiser Permanente MS Clinic Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Advanced Neurology, Fort Collins, Colorado
  - Neurology Associates, PA-Maitland, Maitland, Florida
  - University of South Florida, Morsani College of Medicine, Tampa, Florida
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - University of Kansas Medical Center KUMC - Multiple Sclerosis MS Center, Kansas City, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Dragonfly Research, Wellesley, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - Dent Neurologic Institute, Amherst, New York
  - Columbia University Medical Center-The Neurological Institute of New York, New York, New York
  - University of Rochester Medical Center - URMC, Rochester, New York
  - PMG Research of Piedmont Healthcare, Mooresville, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Premier Neurology P.C., Greer, South Carolina
  - Advanced Neurosciences Institute ANI - Franklin, Franklin, Tennessee
  - Vanderbilt Comprehensive Multiple Sclerosis Center, Nashville, Tennessee
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - MS Center of Greater Washington, Vienna, Virginia
  - Inland Northwest Research LLC, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Griffith University, School of Medicine, Southport, Queensland
- Canada (3):
  - Fraser Health Multiple Sclerosis Clinic, Burnaby, British Columbia
  - Unity Health Toronto/St. Michael's Hospital, Toronto, Ontario
  - Recherche Sepmus Inc., Greenfield Park, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pender MP, Csurhes PA, Smith C, Beagley L, Hooper KD, Raj M, Coulthard A, Burrows SR, Khanna R. Epstein-Barr virus-specific adoptive immunotherapy for progressive multiple sclerosis. Mult Scler. 2014 Oct;20(11):1541-4. doi: 10.1177/1352458514521888. Epub 2014 Feb 3. PMID 24493474
- [Background] Pender MP, Csurhes PA, Burrows JM, Burrows SR. Defective T-cell control of Epstein-Barr virus infection in multiple sclerosis. Clin Transl Immunology. 2017 Jan 20;6(1):e126. doi: 10.1038/cti.2016.87. eCollection 2017 Jan. PMID 28197337
- [Derived] Drosu N, Bjornevik K, Bilodeau PA, Yeh A, Lechner-Scott J, Hawkes CH, Giovannoni G, Levy M. In the era of antiviral trials for MS, the answer lies in the details. Mult Scler Relat Disord. 2024 Feb;82:105444. doi: 10.1016/j.msard.2024.105444. Epub 2024 Jan 12. No abstract available. PMID 38241758
- [Derived] Giovannoni G, Hawkes CH, Lechner-Scott J, Levy M, Yeh EA. Emboldened or not: The potential fall-out of a failed anti-EBV trial in multiple sclerosis. Mult Scler Relat Disord. 2024 Jan;81:105364. doi: 10.1016/j.msard.2023.105364. Epub 2023 Dec 10. No abstract available. PMID 38104476